CLINICAL TRIAL: NCT06286800
Title: Personalized Transcranial Direct Current Stimulation in Stroke Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Timea Hodics, Director, Interventional Neuro-Recovery Program, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00036824
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Transcranial direct current stimulation (ptDCS) (Experimental): TDCS is a noninvasive form of cortical stimulation that uses a battery-powered device. [67] Weak current (0.5-2 mA) will be delivered for up to 20 minutes through surface electrodes which will be positioned using the montage identified as the best in the individual stroke patient during our initial testing session during OT targeting the affected arm.
  Interventions: Device: Transcranial direct current stimulation (tDCS) with OT
- Sham tDCS (Placebo Comparator): Same OT procedure and montage as with the active stimulation but the current will be increased then decreased ramp-like and switched off after 20 seconds instead of the 20 minutes to elicit the same cutaneous sensation as the other stimulation conditions.
  Interventions: Device: Sham tDCS with OT

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) with OT — Weak direct current (0.5-2 mA) will be delivered for up to 20 minutes through surface electrodes which will be positioned using the ptDCS montage. The current will be increased and decreased ramp-like at the beginning and end of the 20-minute stimulation to lessen the itchy/numb skin sensation and decrease the likelihood of an innocuous phosphene-like visual phenomenon. The stimulation will be delivered during the first 20 minutes of occupational therapy targeted to the more affected upper extremity.
  Arms: Personalized Transcranial direct current stimulation (ptDCS)
Device: Sham tDCS with OT — Same procedure and montage as with the active stimulation but the current will be increased then decreased ramp-like and switched off after 20 seconds instead of the 20 minutes to elicit the same cutaneous sensation as the other stimulation conditions. [69] This short length of stimulation is documented to elicit sensations comparable to those of real stimulation. With this procedure, subjects were unable to differentiate between tDCS and sham stimulation in our and other previous studies.
  Arms: Sham tDCS

SUMMARY:
The central objective of this application is to explore the neural substrate of personalized tDCS (ptDCS) and to determine whether the paradigm for each stroke patient can predict the amount of sustained clinical improvement through increased connectivity as measured by a biomarker of plasticity.

DETAILED DESCRIPTION:
This is a randomized, sham controlled double masked parallel group study with optional crossover of chronic (>3mo from stroke onset) ischemic or hemorrhagic stroke patients to test the effect of ptDCS on a cerebral connectivity biomarker of plasticity during stimulation and after 10 treatment of up to 2 mA ptDCS. PtDCS will be performed during the first 20 minutes of occupational therapy targeting the weaker arm compared to sham. Patients will have the option to cross over after the completion of 1-month follow-up and will complete the same procedures with real tDCS if they were in the sham group.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ischemic or hemorrhagic stroke verified by computerized axial tomography or magnetic resonance imaging resulting in hemiparesis (MRC 1-4).
* Age more than 18, Male or Female, All racial and ethnic groups
* Entry into the study >3 months post onset
* Modified Ashworth Scale Score <3 in the involved upper extremity
* Passive range of motion within functional ranges at the shoulder, elbow, wrist and hand
* Able to follow 2 step commands

Exclusion Criteria:

* Patients with history of severe alcohol or drug abuse, psychiatric illnesses like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as unable to follow study instructions).
* Patients with bilateral paresis, or weakness or sensory damage due to peripheral causes (e.g. peripheral nerve injury, muscle or orthopedic injury etc.)
* Patients with severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age,epilepsy or others).
* Patients with unstable cardiac arrhythmia.
* Pregnancy
* Patients with metallic implants in the head, patients with pacemakers, patients with craniotomies, including burr holes who cannot be safely stimulated
* Patients with seizures
* Non-English speaking individuals will only be eligible if they can provide the appropriate translator for all the sessions of the study as no funding is available to pay for such services.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
fMRI functional connectivity biomarker | baseline and 4 weeks
  Task activation, resting state functional connectivity

SECONDARY OUTCOMES:
Wolf Motor Function Test | 4 weeks
  A time-based measurement of upper extremity function of 17 tasks. Shorter performance time is better.
Fugl-Meyer assessment | 4 weeks
  The upper extremity component of Fugl-Meyer test (uFM) is a widely used cumulative numeric rating tool that assesses motor impairment. Range is 0-66, higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Timea Hodics, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States